CLINICAL TRIAL: NCT02983565
Title: The Assessment of Intelligent Oxygen Therapy (iO2T) in Patients With Respiratory Failure on Long-term Oxygen Therapy During Sleep
Brief Title: Intelligent Oxygen Therapy During Sleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 15IC2590
Record Dates: First submitted 2016-11-25; First posted 2016-12-06 (Estimated); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Respiration Failure
Keywords: Long-term oxygen therapy; Intelligent oxygen therapy system; Auto-titrating oxygen system
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participant not aware using iO2T or Fixed flow oxygen
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sleep study on usual long-term oxygen therapy flow rate (No Intervention): Participants will have a sleep study on their usual LTOT flow rate.
- Sleep study on the intelligent oxygen therapy system (Experimental): Participants will have a sleep study on the intelligent oxygen therapy system. This system will supply variable flow oxygen to match a pre-set oxygen saturation target of 93% during sleep.
  Interventions: Device: Intelligent oxygen therapy system (iO2Ts)

INTERVENTIONS:
Device: Intelligent oxygen therapy system (iO2Ts)
  Other Names: Auto-titrating oxygen system
  Arms: Sleep study on the intelligent oxygen therapy system

SUMMARY:
Long-term oxygen therapy improves survival in patients with severe hypoxia. However, some patients despite this oxygen, experience episodes of low oxygen levels (intermittent hypoxia) especially during sleep which may be harmful. In order to overcome this, the investigators have designed an auto-titrating oxygen system (called intelligent oxygen therapy) which automatically adjusts oxygen flow rates to maintain oxygen levels in patients already on oxygen. This study will investigate whether the intelligent oxygen therapy system can prevent intermittent hypoxia during sleep in patients already on long-term oxygen.

DETAILED DESCRIPTION:
Long-term oxygen therapy (LTOT) improves survival in patients with chronic obstructive pulmonary disease (COPD) and severe persistent hypoxia. LTOT is prescribed at a fixed-flow rate with the aim of maintaining a partial pressure of oxygen greater than or equal to 8 kilopascals (kPa). However, a number of studies have demonstrated that patients on home LTOT experience episodes of intermittent hypoxia during rest, activities and especially sleep. Simply increasing the oxygen flow rate at night can relieve this hypoxia but at the expense of hyperoxia with its detrimental effects of hypercapnia and respiratory acidosis. Therefore, a more targeted approach is needed to oxygen delivery. The investigators have devised an auto-titrating oxygen system (intelligent oxygen therapy [iO2Ts]) which delivers variable flow oxygen to maintain a pre-set specific oxygen saturation ( SpO2) target. The system can avoid the dual hazards of hypoxia and hyperoxia and potentially optimise LTOT.

This study will be investigating whether the iO2Ts can reduce intermittent hypoxia during sleep compared to usual fixed flow oxygen in patients on LTOT. Nineteen patients will be recruited to undergo two sleep studies each on two different nights; one on their usual LTOT flow rate and one of the iO2Ts. During both sleep studies, all participants will have full polysomnography, oxygen and transcutaneous carbon dioxide monitoring. The primary outcome will the percentage of time spent with SpO2 < 90% during sleep.

ELIGIBILITY:
Inclusion Criteria:

* On or eligible for long-term oxygen therapy

Exclusion Criteria:

1. Nocturnal use of non-invasive ventilation (NIV) or continuous positive airways pressure (CPAP)
2. A diagnosis of obstructive sleep apnoea
3. A diagnosis of a neuromuscular disease
4. Daytime partial pressure of carbon dioxide > 8.0 kPa
5. Inability to consent for the study
6. Exacerbation of the underlying lung disease or chest infection in the previous 4 weeks
7. Pregnancy
8. Severe co-morbidities
9. Patients with a tracheostomy
10. Long-term oxygen therapy flow rate ≥ 4 litre per minute
11. Inability to understand the English language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
The percentage of time spent with SpO2 <90% during sleep (%) | 10 hours in bed
  The difference in percentage time spent at SpO2 less than 90% during sleeping usual LTOT and iO2T (measured as %)

SECONDARY OUTCOMES:
The percentage of time spent with SpO2 >96% during sleep (%) | 10 hours in bed
  The percentage of time during sleep with an SpO2 value >96% (measured as %)
The mean transcutaneous carbon dioxide level during sleep (measured in kPa) | 10 hours in bed
  Mean level of transcutaneous carbon dioxide level during sleep (measured in kPa)
The peak transcutaneous carbon dioxide level during sleep measures in kPa | 10 hours in bed
  The maximum level of transcutaneous carbon dioxide during sleep (measured in kPa)
The mean sleep SpO2 | 10 hours during sleep
  The mean level of SpO2 during sleep (measured in SpO2 %)
Sleep quality as measured on a visual analogue scale (0 - 100mm). | 10 hours in bed
  The morning after the sleep study, participants will complete a visual analogue scale of their sleep quality. The visual analogue scale is on a A4 paper, it is a straight line of 100mm.
Total Sleep time | 10 hours during sleep
  The total amount of time spent in sleep confirmed by polysomnography (measured in minutes)
Sleep efficiency | 10 hours in bed
  This is the total amount of time the patients actually slept divided by the total time they were in bed (measured as a percentage).

CONTACTS AND LOCATIONS:
Overall Officials: Anita K Simonds, Principal Investigator — Imperial College London
Locations (1):
- Royal Brompton and Harefield NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD.

REFERENCES:
- See also: Completed PhD thesis of M Moghall including results of Intelligent Oxygen therapy during sleep study — https://spiral.imperial.ac.uk/handle/10044/1/59707